CLINICAL TRIAL: NCT04415996
Title: L3/L4 High Velocity Low Amplitude Technique Influence On Baropodometric Pressures In Healthy Young Adults: Randomized Controlled Trial
Brief Title: L3/L4 High Velocity Low Amplitude Technique Influence On Baropodometric Pressures In Healthy Young Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Tecnologia da Saúde do Porto (Other)
Responsible Party: Principal Investigator, Natália Maria Oliveira Campelo, professor, Escola Superior de Tecnologia da Saúde do Porto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: OST1-004
Record Dates: First submitted 2020-05-18; First posted 2020-06-04 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Healthy
Keywords: Lumbar Manipulation; High Velocity Low Amplitude (HVLA) technique; Baropodometry; Osteopathy; Plantar Weight Distribution
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Each participant will pull from a bag within equally number of folded papers with letter A (Intervention Group) and letter B (Control Group) and it will be handled to the investigator.
  The outcome assessors won´t also have any contact with the investigator and participant whilst intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HVLA L3/4 Group (Experimental): In each participant, blind assessors will perform pre-intervention measurements of dislocation of center of pressure (CoP), plantar pressure mean and plantar contact area in a baropodometric pressure platform.
  Next, the investigator will perform the HVLA technique in L3/L4 joint articulation.
  Then, the same measurements before described will be repeated, by the assessors 1 minute after the intervention.
  Interventions: Other: HVLA L3/4
- Control Group (Sham Comparator): In each participant, blind assessors will perform pre-intervention measurements of dislocation of center of pressure (CoP), plantar pressure mean and plantar contact area in a baropodometric pressure platform.
  Next, the investigator will perform a Sham technique. Then, the same measurements before described will be repeated, by the assessors 1 minute after the intervention.
  Interventions: Other: Sham

INTERVENTIONS:
Other: HVLA L3/4 — The participant will be lateral decubitus and the investigator will locate the third lumbar vertebra. Then with one hand the investigator will contact the interspinous space underlying L3 and with the other hand he will take the top leg into flexion until the investigator feels tension in L3/L4 joint. Then he puls the tables´s arm until felling tension in the region to be manipulated. Afterwards the investigator will globally rotate the participant in the horizontal plane and will approach to the L3/L4 joint. With one arm the investigator will contact the deltopectoral groove and with the other one will contact the external iliac fossa. Finally, the investigator will compress and rotate the pelvis and will apply an impulse in a rapid rotation, without losing the parameters with a "body drop" allowed by the flexion of the knees and the contraction of the large pectorals.
  Arms: HVLA L3/4 Group
Other: Sham — The participant will be in lateral decubitus and the top leg and knee will be flexed until the foot reaches the popliteal region of the other leg. There won't be applied any tension in no structure. This intervention will be applied during 20 seconds each side.
  Arms: Control Group

SUMMARY:
In this double-blinded study, the objective is to determine the effects of bilateral High Velocity Low Amplitude (HVLA) technique on L3/L4 joint in baropodometric pressures in 60 healthy young adults.

DETAILED DESCRIPTION:
The postural control it´s a fundamental aspect to understand the human´s capacity to perform activities. These balance is controlled by several mechanisms such as the proprioceptive system of muscles and articulation joints.

It is known that the High Velocity Low Amplitude (HVLA) technique shows biomechanical and neurophysiologic effects.

By saying that, it is importance to understand the effects of the lumbar manipulation on body´s weight distribution. Therefore, there is going to be measure several variables such as center of pressure oscillation , plantar pressure distribution and plantar contact area using a pressure platform.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 18-25 years old;
* Individuals with BMI between 18,5 and 24,9 kg/m2

Exclusion Criteria:

* Pregnancy;
* With the follow conditions: lumbar discal hernia, spondylolisthesis with neurologic influence, narrowing of medullar canal, rheumatic disease, orthopaedic or neurologic conditions such as diminished sensibility, lack or absence of muscular strength, absence of patellar and/or aquilus reflexes;
* History of chirurgical intervention either on lumbar or lower limbs in the past 6 months;
* History of any trauma on the lumbar spine or lower limbs in the past 6 months;
* Any type of treatment on the lumbar in the previous month: that implicates physiotherapy, osteopathy, chiropractic, myofascial treatment, acupuncture or others;
* Medication that affects the vestibular system (dizziness, vertigo and humming)
* Pain during que experimental study;
* Difference between the length of the lower limbs: above 1.5cm;

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline of center of pressure displacement after intervention | Immediately after the intervention
  To obtain the center of pressure displacement measurements, it will be used Emed / CL program. This outcome will be measured either in sagittal plane in anteroposterior direction (x-axis) and in frontal plane in medial-lateral direction (y-axis) The participant will be standing in Emed pressure platform in upright position,with relaxed mouth, upper limbs along the body and feet shoulder-width apart, looking to an object standing 1 meter in front of participant´s eyes during 60 seconds. The Emed/ CL program will determine the This procedure will be repeated 3 times. The participant will rest sited on chair during 30 seconds between each measurements evaluation.

SECONDARY OUTCOMES:
Change from Baseline of plantar pressure mean | Immediately after the intervention
  Plantar pressure mean is measure by Emed / CL program. It´s the average of all pressure values for each measurement, divided by the number of measurements for each sensor. The pressure unit used is Kilopascals (kPa).
  The participant will be standing in Emed pressure platform in upright position,with relaxed mouth, upper limbs along the body and feet shoulder-width apart, looking to an object standing 1 meter in front of participant´s eyes during 60 seconds. This procedure will be repeated 3 times. The participant will rest sited on chair during 30 seconds between each measurements evaluation.
Change from Baseline of plantar contact area | Immediately after the intervention
  Plantar contact area corresponds to the measurement of the contact region of the foot with the platform sensors. It is determined by the sum of the area of all sensors activated within a given region.The plantar contact area unit is cm2 (square centimeters) The participant will be standing in Emed pressure platform in upright position,with relaxed mouth, upper limbs along the body and feet shoulder-width apart, looking to an object standing 1 meter in front of participant´s eyes during 60 seconds. This procedure will be repeated 3 times. The participant will rest sited on chair during 30 seconds between each measurements evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Natália MO Campelo, PhD, Principal Investigator — Escola Superior da Saúde do Porto
Locations (1):
- Escola Superior da Saúde do Porto, Porto, Portugal

REFERENCES:
- [Background] Mendez-Sanchez R, Gonzalez-Iglesias J, Sanchez-Sanchez JL, Puente-Gonzalez AS. Immediate effects of bilateral sacroiliac joint manipulation on plantar pressure distribution in asymptomatic participants. J Altern Complement Med. 2014 Apr;20(4):251-7. doi: 10.1089/acm.2013.0192. Epub 2014 Feb 4. PMID 24494737
- [Background] Gyer G, Michael J, Inklebarger J, Tedla JS. Spinal manipulation therapy: Is it all about the brain? A current review of the neurophysiological effects of manipulation. J Integr Med. 2019 Sep;17(5):328-337. doi: 10.1016/j.joim.2019.05.004. Epub 2019 May 9. PMID 31105036
- [Background] Grassi Dde O, de Souza MZ, Ferrareto SB, Montebelo MI, Guirro EC. Immediate and lasting improvements in weight distribution seen in baropodometry following a high-velocity, low-amplitude thrust manipulation of the sacroiliac joint. Man Ther. 2011 Oct;16(5):495-500. doi: 10.1016/j.math.2011.04.003. Epub 2011 May 14. PMID 21570892
- [Background] Garcia AN, Gondo FL, Costa RA, Cyrillo FN, Silva TM, Costa LC, Costa LO. Effectiveness of the back school and mckenzie techniques in patients with chronic non-specific low back pain: a protocol of a randomised controlled trial. BMC Musculoskelet Disord. 2011 Aug 5;12:179. doi: 10.1186/1471-2474-12-179. PMID 21819594
- [Background] Fagundes Loss J, de Souza da Silva L, Ferreira Miranda I, Groisman S, Santiago Wagner Neto E, Souza C, Tarrago Candotti C. Immediate effects of a lumbar spine manipulation on pain sensitivity and postural control in individuals with nonspecific low back pain: a randomized controlled trial. Chiropr Man Therap. 2020 Jun 3;28(1):25. doi: 10.1186/s12998-020-00316-7. PMID 32487243